CLINICAL TRIAL: NCT04514354
Title: The Influence of Cardiorespiratory Fitness on Firefighter Cardiovascular Health Under Conditions of Heavy Physical Exertion
Brief Title: The Influence of Cardiorespiratory Fitness on Firefighter Cardiovascular Health Under Exercise Conditions
Acronym: FIT & FIRED UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H14-183HH
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases; Post-Exercise Hypotension
Keywords: Firefighters; Post-Exercise Hypotension; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Post-Exercise Hypotension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEST Visit (Experimental): As described in the detailed study description, the GEST Visit included measures of cardiovascular health at Hartford Hospital. These measures included BMI, waist circumference, exhaled carbon monoxide (CO), vascular health (i.e., carotid intimal medial thickness and arterial stiffness), HRV, resting BP, the GEST, and blood draws pre- and post-GEST to obtain SCD and CVD biomarkers.
  Interventions: Behavioral: GEST
- CONTROL Visit (No Intervention): On either Visit 3 or 4, subjects performed the CONTROL Visit. Resting auscultatory blood pressure was measured according to AHA standards. At the conclusion of CONTROL, subjects were fitted for the ABP monitor. Subjects were instructed to proceed with normal activities, not to exercise, and to keep their arm still and extended at their side when each ABP measurement was being taken. Subjects carried a standard journal, recording activities performed during each measurement, any unusual physical or emotional events, and sleep and wake times. The following morning, subjects detached the monitor and returned it that day to the study investigators.

INTERVENTIONS:
Behavioral: GEST — On either Visit 3 or 4, subjects performed a maximal cardiopulmonary GEST following the Balke protocol. Immediately prior to the GEST, the study physician or his designee performed a brief physical examination, in which BP was assessed and all relevant medical information (i.e. medical history, medications, family history) were reviewed. The physician who completed the physical examination remained present during the GEST to monitor the subjects' electrocardiogram (ECG) and other physical signs. After the GEST was completed, the study physician reviewed the ECG for signs of ischemia. Breath-by-breath analysis of expired gases (i.e. oxygen and carbon dioxide) (ParvoMedicsTruneOne® 2400 Metabolic Measurement System, ParvoMedics Inc., Sandy, UT) determined maximal oxygen uptake (VO2max). Heart rate was measured continuously with a 12-lead ECG system and BP was measured by auscultation every 3 minutes during the GEST.
  Arms: GEST Visit

SUMMARY:
Sudden cardiac death (SCD) is the number one cause of on-duty firefighter death. It is most likely to occur in adults who are not physically fit that engage in sudden vigorous exercise. Cardiorespiratory physical fitness (also known as aerobic fitness) is a major heart disease risk factor. In FIT and FIRED UP, the study investigators looked at the influence of cardiorespiratory fitness on blood pressure, heart rate, and other heart markers taken from the blood before and after a vigorous exercise test to maximal effort among firefighters from a local fire department in Connecticut. In addition, the investigators also looked at how lifestyle habits including physical activity, nutrition, stress, and sleep may influence our findings. It was hypothesized that aerobically fit firefighters would show less stress on their heart than unfit firefighters.

DETAILED DESCRIPTION:
The primary purpose of this study was to examine the influence of cardiorespiratory fitness on the acute release of SCD biomarkers and other cardiovascular disease (CVD) risk factors at rest and in response to a bout of maximal physical exertion among 21 firefighters from a local fire department in Connecticut. The study investigators hypothesized that firefighters that are aerobically fit will have lower levels of biomarkers of SCD and a more favorable CVD risk factor profile at rest and in response to a maximal physical effort than firefighters that are not aerobically fit.

FIT and FIRED UP is based on the theoretical foundation of the health belief and social cognitive models of health behavior change which have been shown effective in improving diet and exercise behaviors in firefighters. Specifically, the investigators sought to identify job-specific risk factors for SCD and CVD in firefighters in order to better tailor an intervention that focuses on providing information, reducing barriers to changing unhealthy behaviors, reducing stress, and increasing firefighter efficacy to engage in healthier behaviors.

All eligible members of the fire department were invited to participate in the study. Visit 1 included an orientation health education session at the fire department in which the study investigators delivered a lecture on physical activity and "heart healthy" habits. Interested subjects were able to review the informed consent and questionnaires.

Subjects completed and signed the informed consent at the beginning of Visit 2. This visit consisted of 4 health-related fitness assessments, including sit-up, push-up, flexibility and handgrip tests. Visits 3 and 4 consisted of measures of cardiovascular health at Hartford Hospital and the control visit. The cardiovascular health measures included body mass index (BMI), waist circumference, exhaled carbon monoxide (CO), vascular health (i.e., carotid intimal medial thickness and arterial stiffness), heart rate variability (HRV), resting BP, the maximum graded cardiopulmonary exercise stress test (GEST), and blood draws pre- and post-GEST to obtain SCD and CVD biomarkers. Firefighters were then attached to an ambulatory blood pressure (ABP) monitor and heart rate monitor for 24hr to assess ambulatory BP and HRV, respectively. Of note is that Visits 3 and 4 were conducted in random order so that study investigators could isolate the influence of the GEST on the ambulatory BP response to exercise from the control rest day. Randomization was performed using www.randomization.com. The control visit included measures of resting and ambulatory BP. In addition, subjects completed paper and pencil questionnaires on the topics of physical activity, nutrition, sleep, and mental health at this visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to be full active duty firefighters employed by the local fire department in central Connecticut (CT).
* Subjects confirmed that they were taking the same medication for four weeks prior to Visit 1 and continued taking that medication throughout the duration of the study.

Exclusion Criteria:

* Subjects were excluded from the study if they were not able to comply with all study procedures as described in Visit 1, or in the event of injury or illness that would not enable them to participate.
* If subjects had resting blood pressure readings that were > 160 for systolic blood pressure and/or ≥ 100 mmHg for diastolic blood pressure, they were excluded from the study and referred to their primary care physician for follow up.
* Subjects that were excluded from the study were not penalized in any way by the researchers or the administrators of the local fire department.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Ambulatory Blood Pressure (ABP) | ABP was measured at the conclusion of Visits 3 and 4 during weeks 3 and 4.
  Subjects were attached to an Oscar2 automatic noninvasive ABP monitor (Suntech Medical Instruments Inc., Raleigh, North Carolina, USA) on the nondominant arm to be worn until the next morning. The ABP monitor was programmed to record BP at regular intervals three times per waking hour and two times per sleeping hour.
Change in Resting Blood Pressure | Resting BP was measured during Visits 3 and 4 during weeks 3 and 4.
  Resting BP was measured according to the American Heart Association (AHA) standards using an automated BPTRU monitor (BPTRU Medical Devices, Coquilam, British Columbia, Canada). Subjects were seated for 5 minutes and then BP was measured three times, 1 minute apart in each arm. If the readings obtained were within 5 mmHg, these values were averaged and recorded as resting BP. If these readings did not agree within 5 mmHg, up to three additional readings were taken. If there were three readings obtained that agreed within 5 mmHg, these values were averaged and recorded as resting BP. If after the additional readings were taken and there were not three readings obtained that agree within 5 mmHg, the three closest values were averaged and recorded as resting BP.
Change in Fasted Blood Sampling | The blood sampling occurred at Visit 3 or 4 during the GEST Visit during week 3 or 4.
  The fasting blood sampling occurred prior to and immediately after the GEST and was performed to obtain lipid-lipoprotein profiles and baseline biomarkers associated with cardiovascular disease. A trained phlebotomist collected five tubes of venous blood (52 cc or 3.5 tablespoons) from the antecubital vein of each subject. Serum total cholesterol (mg/dL), triglycerides (mg/dL), high-density lipoprotein cholesterol (HDL-C) (mg/dL), and low-density lipoprotein cholesterol (LDL-C) (mg/dL) were determined by colorimetric enzymatic assays. Serum glucose (mg/dL) was determined by enzymatic/spectrophotometric methods.
Change in Fasted Blood Sampling | The blood sampling occurred at Visit 3 or 4 during the GEST Visit during week 3 or 4.
  The fasting blood sampling occurred prior to and immediately after the GEST and was performed to obtain lipid-lipoprotein profiles and baseline biomarkers associated with cardiovascular disease. A trained phlebotomist collected five tubes of venous blood (52 cc or 3.5 tablespoons) from the antecubital vein of each subject. Serum insulin (uIU/mL) was determined by radioimmunoassay.
Change in Fasted Blood Sampling | The blood sampling occurred at Visit 3 or 4 during the GEST Visit during week 3 or 4.
  The fasting blood sampling occurred prior to and immediately after the GEST and was performed to obtain lipid-lipoprotein profiles and baseline biomarkers associated with cardiovascular disease. A trained phlebotomist collected five tubes of venous blood (52 cc or 3.5 tablespoons) from the antecubital vein of each subject. High sensitivity-C-reactive protein (mg/L) was determined by immunoturbidimetry.
Dietary Intake | The questionnaire was filled out during Visit 3 or 4 at the Control Visit during week 3 or 4.
  Usual dietary and alcohol intake were measured using the National Health and Nutrition Examination Survey (NHANES) semi-quantitative Food-Frequency Questionnaire. The NHANES Food Frequency Questionnaire is a validated tool for measuring dietary intake of both macro- and micro-nutrients based on 127 food items. Subjects were asked to self-report their average daily consumption of 124 food items. The data derived from the Food Frequency Questionnaire were coded and analyzed by members of the National Cancer Institute utilizing Diet*Calc software v1.4.3 (Bethesda, MD) in order to produce daily food frequency estimates of the 127 nutrient and dietary constituents. The Diet*Calc software analyzed Diet History Questionnaire data and generated nutrient and food group intake estimates from the Diet History Questionnaire.
Peak Oxygen Consumption | The GEST took place either during Visit 3 or 4 during week 3 or 4.
  VO2peak was measured by the maximal graded exercise stress test (GEST). The VO2peak test is the gold standard measure of cardiorespiratory fitness.

SECONDARY OUTCOMES:
Health-Related Fitness Assessments | The health-related fitness assessments were performed during study Visit 2 during week 2.
  Subjects performed four health-related fitness assessments. The first assessment was the Flexibility test. All tests were performed with a one-minute rest between tests.
Health-Related Fitness Assessments | The health-related fitness assessments were performed during study Visit 2 during week 2.
  Subjects performed four health-related fitness assessments. The second assessment was the Handgrip Strength test. All tests were performed with a one-minute rest between tests.
Health-Related Fitness Assessments | The health-related fitness assessments were performed during study Visit 2 during week 2.
  Subjects performed four health-related fitness assessments. The third assessment was the Sit-Up test. All tests were performed with a one-minute rest between tests.
Health-Related Fitness Assessments | The health-related fitness assessments were performed during study Visit 2 during week 2.
  Subjects performed four health-related fitness assessments. The fourth assessment was the Push-Up test. All tests were performed with a one-minute rest between tests.
Anthropometrics | Anthropometrics were measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  Height and weight were measured with a calibrated balance beam scale to calculate body mass index (BMI) (kg·m2).
Anthropometrics | Anthropometrics were measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  Waist circumference (cm) was measured at the iliac crest using a non-distensible Guilick tape measure.
Carotid-Intima Media Thickness (cIMT) | CIMT was measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  Subjects rested in the supine position for 5 minutes. CIMT was measured using doppler ultrasound on the carotid arteries at three sites (common, bulb, and internal bilateral). The artery will be imaged using a 5- to 12-MHz multifrequency linear-array transducer attached to a high-resolution ultrasound machine (Terason t3000; Burlington, MA). The image will be digitized and edge detection software (Carotid Analyzer; Medical Imaging Applications, Inc.) will then be used to trace the lumen-intima and intima-medial boundaries of the artery over a 1 minute clip to calculate the average intima-medial thickness at three sites. Mean and maximal distances will be compared to established norms by age, sex/gender, and race/ethnicity.
Change in Arterial Stiffness Assessment | Arterial stiffness was measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  The CPV system (SphygmoCor® CPV Central Blood Pressure/Pulse Wave Velocity System) measured pulse wave velocity (PWV). PWV gives an indication of central arterial parameters. Briefly, the subjects rested in the supine position for 10 minutes. After this rest period, central PWV measures (carotid-femoral), and PWA (radial) were made.
Change in Resting Heart Rate Variability (HRV) | Resting HRV was measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  The resting HRV assessment was performed in a quiet, low-light and temperature-controlled room in the supine position after a 5 min rest period using the GE Case Exercise Testing System (GE Healthcare, Wauwaposa, WI). Following the resting period, electrocardiogram (ECG) RR intervals will be measured in the supine position for 5 min. During these measurements, the subject's breathing frequency was paced at 12 breaths•min-1 with the aid of a metronome.
Change in Ambulatory HRV | Ambulatory HRV was measured during Visit 3 or 4 during the GEST Visit during week 3 or 4.
  Subjects were fitted for a Polar® V800™ HR monitor for the ambulatory HRV assessment for 24 hr. An elastic HR belt was placed below the chest muscles with conductive gel and applied as described by the manufacturer. RR intervals were recorded with a resolution of 1ms and captured by the receptor belt and stored by a wrist watch receiver under free living conditions without controlling for respiratory rate or tidal volume.

CONTACTS AND LOCATIONS:
Overall Officials: Linda S Pescatello, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States